CLINICAL TRIAL: NCT03717532
Title: Blood Flow Restriction Therapy in Patellofemoral Pain Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate/low enrollment
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-01123
Record Dates: First submitted 2018-10-19; First posted 2018-10-24 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Patellopain syndrome with Cuff (Experimental): Patient will be prescribed to 6 weeks of physical therapy with a cuff around the affected leg during exercises
  Interventions: Procedure: Personalized Tourniquet System for Blood Flow Restriction
- Patients with Patellopain syndrome with Placebo Cuff (Placebo Comparator)
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Placebo — Patients will be receiving blood flow restriction therapy with a pressure cuff set to a placebo pressure setting.
  Arms: Patients with Patellopain syndrome with Placebo Cuff
Procedure: Personalized Tourniquet System for Blood Flow Restriction — Patients will be receiving blood flow restriction therapy with a pressure cuff
  Arms: Patients with Patellopain syndrome with Cuff

SUMMARY:
The purpose of this study is to determine the efficacy of blood restriction therapy by comparing increase in muscle mass and strength in patients that receive blood restriction therapy to patients who receive a placebo.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I-II
* Diagnosed with patellofemoral pain syndrome

Exclusion Criteria:

* Patients with confirmed radiographic evidence explaining knee pain
* Legally incompetent or mentally impaired (e.g. minors, Alzheimer's subjects, dementia, etc.)
* Younger than 18 years of age or older than 65
* Any patient considered a vulnerable subject
* Patients with impaired circulation, peripheral vascular compromise, Previous revascularization of the extremity, or severe hypertension
* Patients with Sickle cell anemia or venous thromboembolism
* Patients with Sickle cell anemia or venous thromboembolism
* Patients with cancer or Lymphectomies
* Patients with increased intracranial pressure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Increase in Muscle Mass Measured by Biodex | 6 Weeks
  Biodex dynamometer is used under standard of care to measure the extensor strength of both legs and have bilateral thigh circumference measured
Decrease in Pain measured by Visual Analog Scale (VAS) | 6 Weeks
  100-mm horizontal line anchored at one end with the words "no pain" and at the other end with the words "worst pain imaginable."

CONTACTS AND LOCATIONS:
Overall Officials: Guillen Gonzalez-Lomas, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.